CLINICAL TRIAL: NCT02195024
Title: Cardiac MRI After Replacement of Long Term Implanted PACEmakers by a MRI Conditional Pulse Generator (MRI-rePace)
Brief Title: Cardiac MRI After Pacemaker Replacement
Acronym: MRI-rePACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI changed affiliation not beening allowed to continue the trial in further cooperation. The sub-investigators did not see any option to continue the trial and made the decision to terminate the study.
Sponsor: Dr. Dirk Bastian (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dr. Dirk Bastian, Principal Investigator, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PMUN-DB-001-MRIPM
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Bradycardia; Cardiac Pacemaker; Magnetic Resonance Imaging
Keywords: pacemaker; magnetic resonance imaging; MRI conditional; pacemaker leads
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cardiac MRI group (Active Comparator): • All subjects of the MRI group will undergo a predefined series of magnetic resonance heart scans ≥ six (6) weeks after device exchange
  Interventions: Procedure: cardiac MRI group
- No MRI group (No Intervention): Patients that refuse to undergo cMRI for any reason but accept to attend the trial can be further observed according to the protocol

INTERVENTIONS:
Procedure: cardiac MRI group — • All subjects of the MRI group will undergo a predefined series of magnetic resonance heart scans ≥ six (6) weeks after device exchange
  Arms: cardiac MRI group

SUMMARY:
Aim of this trial is to investigate feasibility of cardiac magnetic resonance imaging (cMRI) in patients with long term implanted coradial leads upgraded to an MRI conditional pacemaker system, to assess MR-image quality and to prove the safety of MRI in this specific population in the short term as well as during long term follow-up.

DETAILED DESCRIPTION:
The trial is designed

1. To investigate the cardiac MRI related adverse event-free rate in patients with long term implanted coradial pacing leads (Fineline-II) after implantable pulse generator (IPG) exchange to a MRI conditional system (short term and long term): Safety.
2. To assess the technical performance of MRI conditional pacemaker systems with long term implanted coradial pacing leads, for cardiac MRI (short term and long term): Effectiveness pacemaker.
3. To assess the image quality (IQ) and the diagnostic value (DV) of the cardiac MRI scans in patients with implanted MRI conditional systems: Effectiveness cardiac MRI.

   2) To evaluate the clinical incidence of MRI procedures in the population of long term implanted pacemaker patients (long term-follow up)

ELIGIBILITY:
Inclusion Criteria:

* Approved clinical indication for pectoral pacemaker exchange (e.g. elective replacement indication (ERI), end of service (EOS))
* Implantation of a CE certified / market released MRI conditional pacemaker (BSCI) consistent of

  * a single or dual chamber MRI conditional pacemaker (BSCI) or
  * Any comparable successor IPG (MRI conditional system, BSCI) compatible with
* Implanted Fineline-II-leads (BSCI), MRI conditional
* Leads electrically intact and with stable and normal function

  * The ascertained lead impedance is between 200 and 1500 Ohm.
  * All pacing capture thresholds (PCT) do not exceed 2.0 V @0.4 or 0.5 ms in pacemaker dependent patients
* Adherence to the MRI conditions of use is given

  * Male or female 18 years or older
  * Understand the nature of the procedure
  * Give written informed consent
  * Able to complete all testing required by the clinical protocol
  * Ability to measure atrial and/or ventricular pacing threshold(s) at 0.4 or 0.5 ms
  * Patient body height greater or equal to 140 cm
  * Pectoral implanted device
  * Subjects who are able and willing to undergo elective cardiac magnetic resonance (MR) scanning without sedation (MRI-group)
  * Subjects who are geographically stable and available for follow-up at the study center for the length of the study

Exclusion Criteria:

* • Non MRI conditional leads implanted

  * Pacing threshold(s) (at 0.4 or 0.5 ms) and/or sensing amplitude(s) and/or impedance(s) are not measurable
  * Meet one or more of the contraindications for MRI including Psychiatric disorders, anxiety, claustrophobia Cardiac disorders that represent a contraindication to MRI
  * Cardiac surgery already scheduled in the next three months
  * Have other medical implants that may interact with MRI, e.g. abandoned implantable cardioverter defibrillator (ICD) leads or pacemaker leads other than MRI conditional, lead extensions, other active medical devices, non-MRI compatible devices, mechanical valve
  * Have other metallic artifacts/components in body that may interact with MRI
  * Subjects for whom a single dose of 1.0 milligram (mg) dexamethasone acetate may be contraindicated
  * Subjects who require a legally authorized representative to obtain consent
  * Subjects who are immediate candidates for an ICD
  * Subjects with medical conditions that preclude the testing required by the protocol or limit study participation
  * Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during this clinical study
  * Being pregnant
  * Have a life expectancy of less than three months
  * Subjects with exclusion criteria required by local law (e.g. age, breastfeeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
safety: cardiac MRI and pacing system related Serious Adverse Device Effects | 3 months after cardiac MRI
  Primary outcome measure 1 (safety):
  * cMRI and pacing system related Serious Adverse Device Effect (SADE) free rate after 3 months.
  * Hypothesis: MRI and pacing system related Serious Adverse Device Effect (SADE) free-Rate is greater than 90% after 3 months.
Effectiveness cardiac MRI: cMRI image quality (IQ) and diagnostic value (DV) | cMRI images done ≥ six (6) weeks after device exchange
  Primary outcome measure 2 (Effectiveness cardiac MRI):
  * cMRI image quality (IQ) and diagnostic value (DV)
  * Hypothesis: cMRI IQ is "acceptable" and clinical use is not adversely affected in ≥ 90% cMRI procedures

SECONDARY OUTCOMES:
cMRI and pacing system related Adverse Device Effect | 1 and 3 months after cardiac MRI
  The proportion of patients with a cMRI and pacing system related Adverse Device Effect (ADE)
Pacemaker performance under/after MRI (short and midterm) - Pacing capture threshold (PCT) rise (atrial and ventricular) | 1 and 3 Months after cardiac MRI
  * The proportion of patients with an atrial or ventricular MRI induced pacing capture threshold rise larger than or equal to 100% voltage safety margin of the measured Pre-MRI pacing threshold at post-MRI interrogation, at 1-month and at 3 month follow- up
  * The proportion of patients with an atrial or ventricular MRI induced pacing threshold rise larger than or equal to 1.0 V @ 0.4 ms or 0.5 ms between pre-MRI and at post-MRI interrogation, 1 month and at 3-month follow-up
Pacemaker performance under/after MRI (short and midterm): atrial or ventricular sensing amplitude | between Pre-MRI evaluation and at post-MRI interrogation at 1-month and at 3-month follow-up after cMRI
  - P and R-wave sensing attenuation:
  o The proportion of patients with an atrial or ventricular amplitude decrease that exceed 50% between Pre-MRI evaluation and at post-MRI interrogation, at 1-month and at 3-month follow-up
- Long term pacing capture threshold rise (atrial and ventricular) | Pre-MRI interrogation and at 2 years follow- up
  * The proportion of patients with an atrial or ventricular MRI induced pacing capture threshold rise larger than or equal to 100% voltage safety margin of the measured Pre-MRI pacing threshold between Pre-MRI interrogation and at 2 years follow- up
  * The proportion of patients with an atrial or ventricular MRI induced pacing capture threshold rise larger than or equal to 1.0 V @ 0.4 ms or 0.5 ms between Pre-MRI interrogation and at 2 years follow- up
- Long term P and R-wave sensing attenuation | between Pre-MRI interrogation and 2 years follow-up
  The proportion of patients with an atrial or ventricular amplitude decrease that exceed 50% between Pre-MRI interrogation and 2 years follow-up
MRI procedures during long term-follow up | during a minimum of 2 years follow-up
  Clinical incidence of MRI procedures during long term-follow up, device performance after repetitive MRI procedures
periprocedural cardiac troponin | pre- and within 3 to 24 hours post-MRI
  Cardiac high sensitive Troponin pre- and post-MRI as marker of thermal injury

OTHER OUTCOMES:
cMRI periprocedural observations / complaints | during cardiac MRI between pre- and post-MRI pacemaker interrogation
  Periprocedural observations / complaints during MRI
  - Time interval: during MRI scanning, between pre- and post-MRI pacemaker interrogation
IPG dysfunction | after cMRI at any follow-up until the end of the trial (minimum 24 months)
  - Any IPG dysfunction (reset, reprogramming, over/undersensing, over-/underpacing, exit-block, loss of capture…), Battery changes

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bastian, MD, Principal Investigator — Paracelsus Medical University Nürnberg
Locations (1):
- Klinikum Nürnberg Süd, Nuremberg, Germany